CLINICAL TRIAL: NCT05315414
Title: An Open, Prospective, Multicenter Investigation to Evaluate the Clinical Outcome of PrimeTaper EV Implant in Extraction Sockets and Healed Ridges - A 5 Year Follow-up
Brief Title: Multicenter Study to Evaluate the Clinical Outcome of PrimeTaper EV Implant in Single Tooth Restorations
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply Sirona Implants and Consumables (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-PT-21-001; NCT05387421 (obsolete NCT alias)
Record Dates: First submitted 2022-03-16; First posted 2022-04-07 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Jaw, Edentulous, Partially
MeSH Terms: conditions — Jaw, Edentulous, Partially

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Single tooth restorations (Experimental): A single, open-label group with patients in need of single tooth restorations will receive PrimeTaper EV implant system with diameters 3.6, 4.2, 4.8, 5.4 mm, and lengths 6.5, 8, 9, 11, 13, 15 and 17 mm.
  Interventions: Device: PrimeTaper EV implant

INTERVENTIONS:
Device: PrimeTaper EV implant — Tapered dental implant developed by Dentsply Sirona

SUMMARY:
The purpose of this study is to evaluate the clinical outcome of implant survival of the PrimeTaper EV implant in single tooth restorations 1 year after permanent restoration.

ELIGIBILITY:
Inclusion Criteria:

* Adult aged 18-75 years.
* Willing and able to sign and date the informed consent form.
* In need of an implant in position 16 to 26 or 36 to 46, and each subject can only receive one implant.
* Deemed by the investigator as likely to present with an initially stable implant situation.
* A stable occlusion, i.e. an opposing natural dentition, a crown, an implant-supported fixed or removable prosthesis, a partial removable prosthesis or a full denture.
* An adjacent tooth (root with natural or artificial crown) or an implant-supported crown mesially and distally. Exemption: If the planned implant is in the first molar position, an edentulous space is accepted distally

Exclusion Criteria:

* Not willing to participate in the clinical investigation or not able to understand the content of the clinical investigation.
* Unlikely to be able to comply with clinical investigation procedures according to investigator's judgement.
* Unable or unwilling to return for follow-up visits for a period of 5 years.
* Known allergy or hypersensitivity to titanium and/or stainless steel.
* Uncontrolled pathological process in the oral cavity, e.g. untreated rampant caries and uncontrolled periodontal disease.
* Uncontrolled para-functional habits, e.g. bruxism.
* Current need of any Guided Bone Regeneration (GBR) procedure in the planned implant area (gap filling at immediate placement and soft tissue grafting are allowed).
* Systemic or local disease or condition that would compromise post-operative healing and/ or osseointegration.
* Immunosuppression, use of corticosteroids, per-os or intravenous bisphosphonate use, or any other medication such as anti-resorptive therapy or monoclonal antibodies that could compromise post-operative healing and/or osseointegration.
* Any other condition that would make the subject unsuitable for participation, including but not limited to;

  * History of radiation therapy in the head and neck region.
  * History of chemotherapy within 5 years prior to surgery.
  * Present alcohol and/or drug abuse.
  * Ongoing psychiatric illness.
  * Current smoking/use of tobacco, including e-cigarettes.
* Any ongoing disease that would make the subject unsuitable for participation, including but not limited to;

  * Recent myocardial infarction (< 3 months*).
  * Recent cerebrovascular accident (< 3 months*).
  * Recent cardiac-valvular prosthesis placement (< 3 months*).
  * Hemorrhagic diathesis.
  * Severe liver dysfunction.
  * Known or suspected current malignancy.
  * Uncontrolled diabetes mellitus.
  * Florid infection.
* Pregnant or breastfeeding females. (Pregnancy tests will be performed as per local requirements).
* Previous enrolment in the present clinical investigation.
* Involvement in the planning and conduct of the clinical investigation (applies to both Dentsply Sirona staff and the clinical investigation site).
* Simultaneous participation in another clinical investigation, or participation in a clinical investigation during the last 6 months that may interfere with the present clinical investigation.

  * < 3 months is a strict exclusion criterion. After 3 month it is up to the investigator to judge whether the subject is considered suitable for participation or not.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2022-05-03 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Implant survival, i.e. number of implants in place counted clinically, 1 year after permanent restoration. | One year post permanent restoration (anticipated average 3 months after implant placement).
  Implant survival rate is a binary variable evaluated clinically, i.e. 'Yes' or 'No' where 'Yes' means that the implant is still in place and 'No' means that the implant is not in place. Any implant that has been removed or lost after implant placement visit will be considered a failure, whatever the reason for removal/loss.

SECONDARY OUTCOMES:
Implant survival, i.e. number of implants in place counted clinically, 2, 3, 4 and 5 years after permanent restoration. | 2, 3, 4 and 5 years post permanent restoration (anticipated average 3 months after implant placement).
  Implant survival rate is a binary variable evaluated clinically, i.e. 'Yes' or 'No' where 'Yes' means that the implant is still in place and 'No' means that the implant is not in place. Any implant that has been removed or lost after implant placement visit will be considered a failure, whatever the reason for removal/loss.
Change of implant stability quotient value (ISQ) between implant placement and permanent restoration. | From date of implant placement (anticipated average 1 month after inclusion) to date of permanent restoration (anticipated average 3 months after implant placement).
  Implant stability will be evaluated through ISQ value using Resonance Frequency Analysis (RFA). The stability is presented as an ISQ value. The higher the ISQ value the higher the stability. Recorded as a numeric value (1-100).
Maximum insertion torque value for each implant at implant placement. | At date of implant placement (anticipated average 1 month after inclusion).
  Maximum insertion torque value (ITV), based on ITV curve, measured in Ncm.
Final insertion torque value for each implant at implant placement. | At date of implant placement (anticipated average 1 month after inclusion).
  Final insertion torque value (ITV), based on ITV curve, measured in Ncm.
Investigator questionnaire for each investigational medical device after implant placement. | Immediately after implant placement (anticipated average 1 month after inclusion).
  Numerical scale 1-10, where 1 = totally disagree with the statement, and 10 = totally agree with the statement. Statements to be evaluated by the surgeon: "The implant was guided into the prepared osteotomy", "The implant followed the prepared osteotomy", "The implant has a good primary stability", "The drilling protocol is easy to use", "The implant has efficient cutting properties". Each statement will be evaluated separately.
Implant success, i.e., number of implants documented as successful at 1, 2, 3 and 5 years after permanent restoration. | 1, 2, 3 and 5 years post permanent restoration (anticipated average 3 months after implant placement).
  Successful implants counted, i.e. 'Yes' or 'No'. An implant will be considered successful if all of the following criteria are fulfilled:
  1. Implant in place.
  2. Lack of evidence of peri-implant radiolucency in X-ray.
  3. Less than 1mm vertical bone loss during first year after loading with permanent restoration and 0,2mm annually thereafter.
  4. Absence of persistent and/or irreversible signs and symptoms such as pain, infections, neuropathies, paresthesia, or violation of the mandibular canal.
Change of marginal bone level up to 5 years post permanent restoration compared to permanent restoration. | At permanent restoration (anticipated average 3 months after implant placement) and 1, 2, 3 and 5 years post permanent restoration.
  MBL changes determined from radiographs, expressed as the distance from the implant reference point to the most coronal bone-to-implant contact on the mesial and distal side of the implant. The average will be calculated and compared for each evaluation period.
Change of probing pocket depth (PPD) in mm between permanent restoration, and 6 months, 1, 2, 3, 4 and 5 years after permanent restoration. | At permanent restoration (anticipated average 3 months after implant placement) and 6 months, 1, 2, 3, 4 and 5 years post permanent restoration.
  Probing Pocket Depth (PPD) measured as the distance from the mucosal margin to the bottom of the probe-able pocket in mm.
Presence of bleeding on probing (BoP), at permanent restoration, and 6 months, 1, 2, 3, 4 and 5 years after permanent restoration. | At permanent restoration (anticipated average 3 months after implant placement) and 6 months, 1, 2, 3, 4 and 5 years post permanent restoration.
  Bleeding on Probing (BoP) recorded as presence or absence of bleeding when probing to the bottom of the pocket.
Presence of plaque at 6 months, 1, 2, 3, 4 and 5 years after permanent restoration. | 6 months, 1, 2, 3, 4 and 5 years post permanent restoration (anticipated average 3 months after implant placement).
  Plaque recorded as presence or absence of plaque by visual inspection on four surfaces at each implant site.
Occurrence of Adverse Events, Adverse Device Effects, and Device Deficiencies during the clinical investigation. | Up to 5 years after permanent restoration (anticipated average 3 months after implant placement).
  Adverse Events, Adverse Device Effects, and Device Deficiencies spontaneously reported, and collection at each clinical investigation visit.

CONTACTS AND LOCATIONS:
Overall Officials: Andy Temmerman, Prof., Principal Investigator — KU Leuven
Locations (5):
- University of Iowa, Iowa City, Iowa, United States
- Catholic University of Leuven, Leuven, Belgium
- Dental practice Dr Mischa Krebs, Alzey, Germany
- Studio Toia, Busto Arsizio, Italy
- Dr.F.L.Guljé, De Mondhoek, Apeldoorn, Netherlands